CLINICAL TRIAL: NCT06285097
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETIC, PHARMACODYNAMIC, AND ANTITUMOR ACTIVITY OF PF-07820435 AS MONOTHERAPY AND IN COMBINATION IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study of PF-07820435 as a Single Agent and in Combination in Participants With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated for strategic business reasons; the decision was not based on any safety and/or efficacy concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C5391001; NCT06285097 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-01-23; First posted 2024-02-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms; Non-small-cell Lung Cancer; Melanoma; Squamous Cell Carcinoma of the Head and Neck; Renal Cell Carcinoma; Urothelial Carcinoma; Colorectal Carcinoma; Ovarian Carcinoma
Keywords: Sasanlimab; anti-Programmed death receptor-1 (PD-1); solid tumor; immunotherapy
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Renal Cell; Carcinoma, Transitional Cell; Colorectal Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Monotherapy dose escalation (Part 1A) (Experimental): Participants will receive PF-07820435 orally at the prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07820435
- Combination dose escalation (Part 1B) (Experimental): Participants will receive PF-07820435 orally at the prescribed dose and frequency, in combination with sasanlimab (subcutaneous injection) at a fixed dose once every 4 weeks in 28-day cycles
  Interventions: Drug: PF-07820435; Biological: Sasanlimab
- Expansion (Part 2) - Tumor specific Arm A (Experimental): Participants will receive PF-07820435 orally at the prescribed dose and frequency in combination with sasanlimab SC once every 4 weeks in 28-day cycles
  Interventions: Drug: PF-07820435; Biological: Sasanlimab
- Expansion (Part 2) - Tumor specific Arm B (Experimental): Participants will receive PF-07820435 orally at the prescribed dose and frequency in combination with sasanlimab SC once every 4 weeks in 28-day cycles
  Interventions: Drug: PF-07820435; Biological: Sasanlimab
- Expansion (Part 2) - Arm C (Experimental): Participants will receive PF-07820435 orally at the prescribed dose and frequency in 28-day cycles
  Interventions: Drug: PF-07820435

INTERVENTIONS:
Drug: PF-07820435 — immune agonist
Biological: Sasanlimab — A monoclonal antibody that blocks the interaction between PD-1 and PD-L1/L2
  Arms: Combination dose escalation (Part 1B); Expansion (Part 2) - Tumor specific Arm A; Expansion (Part 2) - Tumor specific Arm B

SUMMARY:
This study aims to evaluate the safety, and early signals of anti-tumor activity of PF-07820435 when administered alone (Part 1A) or in combination with sasanlimab (Part 1B; Part 2) in patients with selected advanced or metastatic solid tumors. Part 1 will be dose-finding and Part 2 of the study will further evaluate PF-07820435 at the recommended dose for combination expansion in patients with selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of advanced, unresectable, and/or metastatic or relapsed/refractory solid tumor
* Part 1A: Participants with solid tumors where anti-PD-(L)1 is an established treatment. Participants must have progressed on or following prior anti-PD-(L)1 therapy if approved, available, tolerable, and eligible
* Part 1B: Participants either meeting Part 1A criterion, or participants with "cold" solid tumors where anti-PD-(L)1 therapy is not an established treatment
* Part 2: Participants with NSCLC (Arm A) must have received platinum-based chemotherapy and anti-PD-(L)1 or have intolerability to or refusal of standard therapies. NSCLC participants with known activating mutation(s) must also have received prior approved and available targeted therapy(ies) for the associated mutation(s) or have intolerability or documented refusal of these therapies. Participants with UC (Arm B) must have received prior platinum-based chemotherapy, anti-PD-(L)1 therapy, or enfortumab vedotin, or have documented intolerability or refusal of the standard therapy(ies). Additional cohort indication(s) or dose regimens may be added and defined based on emerging data
* At least 1 measurable lesion based on RECIST 1.1 that has not been previously irradiated (Part 1 exceptions permitted after review and approval)
* Able to provide pre-treatment (and optional on-treatment) tumor tissue

Exclusion Criteria:

* Active or history of clinically significant gastrointestinal disease and other conditions that are unresolved or pose a risk to study treatment or procedures
* Active or history of pneumonitis/interstitial lung disease, pulmonary fibrosis requiring treatment with systemic steroid therapy
* Active or history of clinically significant autoimmune disease or other medical condition that required chronic systemic immunosuppressive therapy within recent 2 years
* History of severe immune-mediated adverse event or cytokine release syndrome that was considered related to prior immune modulatory therapy that required immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Number of patients with dose limiting toxicities (DLTs) in dose escalation (Part 1A and Part 1B) | Baseline through 28 days after first dose
  DLT rate estimated based on data from DLT-evaluable participants during the DLT evaluation period
Number of patients with adverse events (AEs) | Baseline through up to 2 years
  Characterized by type, frequency, severity (CTCAE v5; CRS by ASTCT), timing, seriousness, and relationship to study drug(s)
Number of patients with clinically significant lab abnormalities | Baseline through up to 2 years
  Characterized by type, frequency, severity (CTCAE v5), and timing
Objective response rate (ORR) in Part 2 Expansion | Baseline through 2 years or disease progression
  Tumor response as assessed using RECIST 1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) in dose escalation (Part 1A and Part 1B) | Baseline through 2 years or disease progression
  Tumor response as assessed by RECIST 1.1
Duration of tumor response | Baseline through 2 years or disease progression
  Tumor response as assessed by RECIST 1.1
Progression free survival (PFS) | Baseline through 2 years or disease progression
  Tumor response as assessed by RECIST 1.1
Cmax (maximum concentration) of PF-07820435 and its active metabolite | Serial timepoints following the first dose (Day 1), second dose (Day 8), and third dose (Day 15) of the first cycle (each cycle is 28 days); and Day 1 (dosing) of Cycle 2 and Day 1 (dosing) of Cycle 3.
  Single and multiple dose PK parameters of PF-07820435 and its active metabolite
Tmax (time to maximal plasma concentration) of PF-07820435 and its active metabolite | Serial timepoints following the first dose (Day 1), second dose (Day 8), and third dose (Day 15) of the first cycle (each cycle is 28 days); and Day 1 (dosing) of Cycle 2 and Day 1 (dosing) of Cycle 3.
  Single and multiple dose PK parameters of PF-07820435 and its active metabolite
AUClast (area under the curve from time 0 to the last measurable timepoint) of PF-07820435 and its active metabolite | Serial timepoints following the first dose (Day 1), second dose (Day 8), and third dose (Day 15) of the first cycle (each cycle is 28 days); and Day 1 (dosing) of Cycle 2 and Day 1 (dosing) of Cycle 3.
  Single and multiple dose PK parameters of PF-07820435 and its active metabolite
Cmin (minimum concentration) of PF-07820435 and its active metabolite after multiple dosing only | Serial timepoints following the first dose (Day 1), second dose (Day 8), and third dose (Day 15) of the first cycle (each cycle is 28 days); and Day 1 (dosing) of Cycle 2 and Day 1 (dosing) of Cycle 3.
  Multiple dose PK parameters of PF-07820435 and its active metabolite
Change from baseline of immune markers within biopsied tumor tissue | Baseline through about 6 weeks after first dose
  Change in CD8 immune marker will be analyzed
Pre-dose trough concentrations of sasanlimab (Part 1B and Part 2) | Day 1 (pre-dose) of each cycle (28 days) for the first 3 cycles, then Day 1 on every 3rd cycle until 2 years or disease progression
  Single and multiple dose PK parameters of sasanlimab
Incidence and titers of ADA and NAb against sasanlimab (Part 1B and Part 2) | Day 1 (pre-dose) of each cycle (28 days) for the first 3 cycles, then Day 1 on every 3rd cycle until 2 years or disease progression
  Immunogenicity assessment
Cmax of PF-07820435 and its active metabolite under fasted and fed conditions (Part 2 subset) subset of participants in Part 2 | On Day 1 (first dose) and Day 15 (third dose): Pre-dose, 0.5 hour (h), 1h, 2h, 4h, 6h, and 24h post dose.
  The analysis applies to Part 2 Food Effect Subset only
Tmax of PF-07820435 and its active metabolite under fasted and fed conditions (Part 2 subset) subset of participants in Part 2 | On Day 1 (first dose) and Day 15 (third dose): Pre-dose, 0.5 hour (h), 1h, 2h, 4h, 6h, and 24h post dose.
  The analysis applies to Part 2 Food Effect Subset only
AUC of PF-07820435 and its active metabolite under fasted and fed conditions (Part 2 subset) subset of participants in Part 2 | On Day 1 (first dose) and Day 15 (third dose): Pre-dose, 0.5 hour (h), 1h, 2h, 4h, 6h, and 24h post dose.
  The analysis applies to Part 2 Food Effect Subset only

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (6):
  - Florida Cancer Specialists Sarasota Drug Development Unit, Sarasota, Florida
  - Corewell Health (reference non-engagement letter), Grand Rapids, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tristar Centennial Medical Center, Nashville, Tennessee
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
- Puerto Rico (2):
  - Hospital Oncologico Dr. Isaac Gonzalez-Martinez, Rio Piedras
  - Pan American Center for Oncology Trials, LLC, Rio Piedras

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5391001